CLINICAL TRIAL: NCT06503601
Title: The Impact of Genetic Polymorphism on the Echocardiographic Parameters and Cardiac Fibrosis Markers in Response to Empagliflozin Treatment Among Patients With Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ruwan Mokhtar, Teaching Assistant, Ain Shams University
Other Study IDs: rec#264
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; genetic polymorphism; cardiac fibrosis markers; empagliflozin; echocardiographic parameters
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Responders to empagliflozin: Heart failure patients who showed response to empagliflozin
- Non responders to empagliflozin: Heart failure patients who showed no response to empagliflozin

SUMMARY:
It is important to assess the implications of genetic variants of the TGF-β1 gene in patients with HFrEF and the association of this polymorphism with treatment response to SGLT2I. Therefore, by correlating the pharmacogenetics hand in hand with the mechanistic markers involved in the pathogenesis of HF, this can aid in the development of individualized, therapeutic strategies and improve the patient's drug response.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of morbidity and mortality worldwide. According to the American heart association (AHA) over 19.1 million deaths worldwide in 2020 were attributed to CVD. Heart failure (HF) is considered one of the most frequent causes of hospitalization and the final stage of many heart disorders. It is associated with high rates of morbidity and mortality. Heart failure (HF) affects more than 5.8 million people in the USA and over 23 million people worldwide, making it a serious public health issue. According to the 2022 guidelines of American heart association (AHA) a variety of non-pharmacologic and pharmacologic are available to treat heart failure (HF) to prevent or reverse its symptoms. Nonpharmacologic treatments may involve dietary sodium and fluid restriction, proper physical activity, and attention to weight gain depending on the illness's severity. Pharmacologic treatments include the use of diuretics, vasodilators, inotropic agents, anticoagulants, beta blockers, angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), calcium channel blockers (CCBs), digoxin, nitrates, B-type natriuretic peptides (BNPs), I(f) inhibitors, angiotensin receptor-neprilysin inhibitors (ARNIs), soluble guanylate cyclase stimulators, sodium-glucose cotransporter-2 inhibitors (SGLT2Is), and mineralocorticoid receptor antagonists (MRAs). Recent study has shown that SGLT2I not only lowers blood sugar levels but also protects the kidney and heart, which can dramatically lower cardiovascular events, stall the advancement of renal failure, significantly raise patient quality of life, and lower medical costs for families and society. A study showed that Empagliflozin has cardio-renal protective effects as it reduced inflammatory and fibrotic markers, such as NF-κB, TGF-β1, and improved fibrosis. However, it was found that the variation in treatment response with SGLT2I may be due to the genetic polymorphism of TGF-β1 since this polymorphism may influence its expression. Therefore, it is important to assess the implications of genetic variants of the TGF-β1 gene in patients with HFrEF and the association of this polymorphism with treatment response to SGLT2I. Therefore, by correlating the pharmacogenetics hand in hand with the mechanistic markers involved in the pathogenesis of HF, this can aid in the development of individualized, therapeutic strategies and improve the patient's drug response.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients NYHA class II to IV.
* Treatment with beta blockers, MRAs, ACEIs in addition to empagliflozin.
* Age of 18 years to 80 years.
* Written informed consent of the subject to participate in the study.

Exclusion Criteria:

* Contraindication to empagliflozin: pregnancy, hypersensitivity, and severe renal impairment.
* CABG or valve surgery within 3 months.
* Mild-to-severe valvular stenosis or severe (grade III/IV) valvular regurgitation
* Pregnant or nursing women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients treated with empagliflozin
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphism and echocardiographic parameters | 3-6 months
  To detect association between a TGFβ1 gene polymorphism variants and echocardiographic outcome of patients with HFrEF in response to empagliflozin.

SECONDARY OUTCOMES:
Cardiac fibrosis biochemical markers | 3-6 months
  • To detect association between serum TGFβ1, MMP-2 and TNF-α levels (cardiac fibrosis biochemical marker) and echocardiographic parameters of patients with HFrEF in response to empagliflozin

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided